CLINICAL TRIAL: NCT04830956
Title: Evaluation of Comfort in Subjects With Moderate Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DEJ475-E004
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Sequence 1 (Experimental): FID123238 in 4 specification levels (minimum, moderate, moderate plus, maximum) and Systane hydration applied to the ocular surface in 1 of 5 randomized sequences. 1 application per product.
  Interventions: Other: FID123238; Other: Systane Hydration
- Sequence 2 (Experimental): FID123238 in 4 specification levels (minimum, moderate, moderate plus, maximum) and Systane hydration applied to the ocular surface in 1 of 5 randomized sequences. 1 application per product.
  Interventions: Other: FID123238; Other: Systane Hydration
- Sequence 3 (Experimental): FID123238 in 4 specification levels (minimum, moderate, moderate plus, maximum) and Systane hydration applied to the ocular surface in 1 of 5 randomized sequences. 1 application per product.
  Interventions: Other: FID123238; Other: Systane Hydration
- Sequence 4 (Experimental): FID123238 in 4 specification levels (minimum, moderate, moderate plus, maximum) and Systane hydration applied to the ocular surface in 1 of 5 randomized sequences. 1 application per product.
  Interventions: Other: FID123238; Other: Systane Hydration
- Sequence 5 (Experimental): FID123238 in 4 specification levels (minimum, moderate, moderate plus, maximum) and Systane hydration applied to the ocular surface in 1 of 5 randomized sequences. 1 application per product.
  Interventions: Other: FID123238; Other: Systane Hydration

INTERVENTIONS:
Other: FID123238 — Lubricant applied to the ocular surface
Other: Systane Hydration — Drops applied to the ocular surface

SUMMARY:
The purpose of this study is to evaluate the comfort of an ocular lubricant in dry eye subjects. This study will be conducted in Canada and Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an information consent letter
* Willing and able to follow instructions and maintain the appointment schedule
* Has dry eye symptoms

Key Exclusion Criteria:

* Has suffered any ocular injury to either eye in the past 12 weeks
* Is pregnant or lactating at the time of enrollment

Other protocol-specified inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in comfort rating | Baseline, up to 12 Hours (Day 1, each product)
  A visual analogue scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (1):
- Alcon Investigator 8169, Carlton, Victoria, Australia